CLINICAL TRIAL: NCT06785493
Title: A Retrospective Analysis on the Clinical Efficacy and Influence Factors of Individualized Treatment of Ustekinumab in Patients With Crohn's Disease
Brief Title: The Clinical Efficacy and Influence Factors of Individualized Treatment of Ustekinumab in Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-201
Record Dates: First submitted 2025-01-13; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: IBD (Inflammatory Bowel Disease)
Keywords: Ustekinumab; Individualized treatment; Clinical efficacy; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Optimized Treatment (OPT) — After the first sufficient intravenous infusion of UST (6 mg/kg), the patient's response was assessed based on PRO2 at week 8, and an individualized treatment plan was developed. At week 8, the patients with incomplete response of PRO2 (a decline of PRO2 was less than 50% from baseline or still in moderate to severe active phase of PRO2) were given one or more UST intravenous re-induction (6 mg/kg) every 4 or 6 weeks.

SUMMARY:
The loss of response rate of ustekinumab(UST) is high, and the specific mechanism has not yet been elucidated. Our study aimed to retrospectively analyze the clinical efficacy and influence factors of individualized treatment of ustekinumab (UST) in patients with Crohn's disease (CD).

DETAILED DESCRIPTION:
Interleukin (IL-12) and interleukin (IL-23) co-contain the P40 subunit, and ustekinumab (UST) is a fully humanized IgG1 monoclonal antibody that targets the P40 subunit. The conventional regimen of UST in the treatment of Crohn's disease is that after the first sufficient dose (6 mg/kg) of intravenous infusion, 90 mg UST is injected subcutaneously at the 8th week according to the patient's response, and maintenance therapy is given every 8 or 12 weeks. However, data from real-world studies suggest that the clinical efficacy of treating CD with the conventional UST regimen is less than ideal.Our study aimed to retrospectively analyze the clinical efficacy and influence factors of individualized treatment of ustekinumab in patients with Crohn's disease .

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with moderate to severe Crohn's disease
2. Receiving treatment with ustekinumab

Exclusion Criteria:

1. Combined with other autoimmune diseases (such as systemic lupus erythematosus, Sjogren's syndrome, etc.), malignant tumors, or severe cardiovascular and cerebrovascular diseases
2. Merge active tuberculosis or severe infection
3. Liver and kidney dysfunction
4. Pregnancy or lactation period
5. Combination therapy with hormones, immunosuppressants, small molecule drugs, or other biological agents
6. Clinical data missing ≥ 30% or lost to follow-up during the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inflammatory bowel disease (IBD) is a chronic inflammatory disease involving the digestive tract, including two clinical phenotypes: Crohn's disease (CD) and ulcerative colitis (UC).
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
The endoscopic efficacy of ustekinumab treatment at week 36 | at week 36
  Simplified Crohn's Disease Endoscopic Score (SES-CD) was employed to evaluate the degree of intestinal inflammation of CD patients.Intestinal inflammation was assessed as mild (3-6 points) , moderate (7-15 points) , and severe (≥16 points) .
The clinical efficacy of ustekinumab treatment at week 36 | at week 36
  Harvey-Bradshaw Index (HBI) was applied to assess the clinical activity of CD patients.HBI is divided into mild (5-7 points), moderate (8-16 points), and severe (≥ 17 points).

SECONDARY OUTCOMES:
influencing factors | at week 36
  At week 36, analyze the influencing factors of clinical remission rate(HBI≤ 4 points) .
influencing factors | at week 36
  At week 36, analyze the influencing factors of endoscopic remission rate(SES-CD ≤ 2 points, or no ulcers).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No